CLINICAL TRIAL: NCT00848965
Title: A Randomised, Double Blind, Placebo Controlled, 4 Period, Incomplete Block, Crossover Study to Assess the Dose-response Curve of Intranasal Fluticasone Propionate (25, 50, 100 and 200 μg, Once Daily for 8 Days) in the Vienna Challenge Chamber for the Purpose of Investigating the Sensitivity
Brief Title: A Randomised, Double Blind, Placebo Controlled, 4 Period, Incomplete Block, Crossover Study Assessing the Dose-response Curve of Fluticasone Propionate in an Antigen Challenge Chamber
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 110341; 781 IIa
Record Dates: First submitted 2009-02-12; First posted 2009-02-23 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2011-02

CONDITIONS: Rhinitis, Allergic, Perennial; Allergic Rhinitis
Keywords: fluticasone propionate; Vienna Challenge Chamber; glucocorticosteroids; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Fluticasone propionate 25ug (Experimental)
  Interventions: Drug: Fluticasone propionate
- Fluticason propionate 50ug (Experimental)
  Interventions: Drug: Fluticasone propionate
- Fluticasone propionate 100ug (Experimental)
  Interventions: Drug: Fluticasone propionate
- Flutciasone propionate 200ug (Experimental)
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Fluticasone propionate — Corticosteriod, with anti-inflammatory effects
  Arms: Flutciasone propionate 200ug; Fluticason propionate 50ug; Fluticasone propionate 100ug; Fluticasone propionate 25ug
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This is a single-centre, randomised, double-blind, four-period, incomplete block, crossover study, with 8 days repeat dosing of intranasal Fluticasone Propionate (25, 50, 100, 200ug) and/or placebo in the Vienna Challenge Chamber in subjects with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy with the exception of seasonal allergic rhinitis. Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* Males and females who are aged between 18 and 65 years of age.

A female is eligible to enter and participate in the study if she is of:

1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who is post menopausal. For the purposes of this study, post menopausal is defined as 1 year without menses (FSH/LH will be also tested to confirm menopausal status); or
2. Child bearing potential, has a negative pregnancy test (urine) at entry, and agrees to one of the following acceptable contraceptive methods when used consistently and correctly (i.e., in accordance with the approved product label and the instructions of a physician for the duration of the study - screening visit to follow-up contact):

   * Complete abstinence from intercourse from the first visit, throughout the trial and for a minimum of 7 days after the completion of the trial; or
   * Male partner was sterile prior to the female subject's entry into the study, or
   * Implants of levonorgestrel inserted for at least 1 month prior to the study
   * Injectable progestogen administered for at least 1 month prior to the study
   * Oral contraceptive (combined or progestogen only) administered for a least one monthly cycle prior to study medication administration; or
   * The contraceptive transdermal patch, such as norelgestromin / ethinyl estradiol transdermal system (if the subject is less than 89kg); or
   * Double-barrier method - spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a spermicide and female diaphragm .
   * Condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; or
   * An intrauterine device (IUD) or intrauterine system (IUS), inserted by a qualified physician,
   * Subjects who are current non-smokers, who have not used any inhaled tobacco products (snuff is permitted) in the 12 month period preceding the screening visit and who have a pack history of less than 10 pack years.

Pack years = Number of cigarettes per day x Number of years smoked 20

* They exhibit a moderate response to up to 1500 grass pollen grains/m3 after 2 hours in the Vienna Challenge Chamber, which is defined as a nasal symptom score of at least 6. (Nasal symptom score is the sum of nasal obstruction, rhinorrhoea, nasal itch and sneeze, each of which are scored on a scale from 0 to 3)
* They have a positive skin prick test (wheal ³ 4mm) for grass pollen at or within the 12 months preceding the screening visit.
* They have a positive RAST (Radioallergosorbent Test) (³ class 2) for grass pollen at or within the 12 months preceding the screening visit.
* They have a TNSS score (Total Nasal Symptom Score)of less than 3 and a score of no more than 1 for any single symptom of the TNSS prior to the screening allergen challenge.
* There are no conditions or factors that would make the subject unlikely to be able to stay in the trial
* Able to provide written informed consent.
* The subject is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.
* Demonstrated ability to use the intranasal device in a satisfactory and repeatable manner.

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigations, the principle investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 150 mmHg or a diastolic pressure above 90 mmHg unless the Investigator confirms that it is satisfactory for their age.
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
* Pregnant or nursing females.
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception as outlined (Inclusion Criteria 2)
* On examination the subject is found to have any structural nasal abnormalities or nasal polyposis, a history of frequent nosebleeds, recent nasal surgery or recent (within 2 weeks) or ongoing upper respiratory tract infection which in the Responsible Physician's opinion renders the subject unsuitable for participation in the study.
* Any respiratory disease other than mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function.
* The subject is likely to be unable to abstain from salbutamol use for 8 hours before a challenge.
* The subject has a screening QTcB value >450msec (based on single or average QTc value of triplicate ECGs obtained over a brief recording period), PQ interval outside the range 120 to 200msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T-wave). In addition subjects will be excluded if they have a history of atrial or ventricular arrhythmia.
* The subject has a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* The subject has taken prescription or non-prescription drugs, within 7 days prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* History of alcohol/drug abuse or dependence within 12 months of the study. Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine).
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has donated a unit of blood (450 mL) within the previous 16 weeks or intends to donate within 16 weeks after completing the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has tested positive for HIV antibodies (if tested according to site Standard Operating Procedures).
* The subject has a positive pre-study urine drug/ urine alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids (THC) and Benzodiazepines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) were randomized to receive treatment in one of five sequences in four study periods: ABCD, EABC, DEAB, CDEA, BCDE (A, Placebo; B, fluticasone propionate [FP] 25 micrograms [µg]: C, FP 50 µg; D, FP 100 µg; E, FP 200 µg). One par. randomized to ABCD withdrew due to an adverse event; one par. randomized to EABC withdrew consent.
Groups:
- Placebo/FP 25, 50, 100, 200 µg: Participants received placebo/fluticasone propionate (FP) in a dose of 25, 50, 100, and 200 micrograms (µg) once daily as 1 nasal spray into each nostril from 2 separate devices for 8 days each, in a crossover design. Treatment was given in one of five sequences in Periods 1, 2, 3, and 4 (with a minimum of a 14-day washout period between treatments): ABCD, EABC, DEAB, CDEA, and BCDE (A, Placebo; B, FP 25 µg: C, FP 50 µg; D, FP 100 µg; E, FP 200 µg). On Day 8 of each treatment period (1 hour post-dose), participants entered the Vienna Challenge Chamber (VCC) for a 4-hour period, and the assessments were conducted 2-5 hours post-dose. All participants attended a follow-up visit within 2 to 4 weeks after their final dose, and the overall duration for participation in the study (screening to follow-up) did not exceed 158 days.
Period: Overall Study
Arm/Group | Placebo/FP 25, 50, 100, 200 µg
Started | 59
Completed | 57
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Placebo/FP 25, 50, 100, 200 µg
Number analyzed (Participants) | 59
Age Continuous [Mean (Standard Deviation); unit: Years] | 27.2 (5.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese/East Asian Heritage (EAH)/South EAH | 1
  White | 58

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean Total Nasal Symptom Score (TNSS) at 2-5 Hours Post-dose (1-4 Hours Post-start of Challenge [PSC]) in the Vienna Challenge Chamber (VCC)
Description: The TNSS (score of 0-12), defined as the sum of the symptom scores for nasal obstruction, rhinorrhea, nasal itch, and sneeze (each scored on 0-3 scale [0=none, 1=mild, 2=moderate, 3=severe]) was measured at pre-challenge, and then every 15 minutes from 0.25 to 4 hours PSC. In the VCC, aerosolized allergen is administered in a sealed chamber to evaluate the efficacy of antihistamines/other treatments. Weighted mean TNSS was calculated by dividing the value of the area under the response time curve between 1 and 4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each study period (Periods 1-4); up to Day 158
Population: All Subjects Population: all participants randomized to receive at least one dose of study treatment. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Placebo: Participants received identical placebo once daily as 1 nasal spray into each nostril from separate devices for 8 days
- 25 µg FP: Participants received FP in a dose of 25 µg once daily as 1 nasal spray into each nostril from separate devices for 8 days
- 50 µg FP: Participants received FP in a dose of 50 µg once daily as 1 nasal spray into each nostril from separate devices for 8 days
- 100 µg FP: Participants received FP in a dose of 100 µg once daily as 1 nasal spray into each nostril from separate devices for 8 days
- 200 µg FP: Participants received FP in a dose of 200 µg once daily as 1 nasal spray into each nostril from separate devices for 8 days
Arm/Group | Placebo | 25 µg FP | 50 µg FP | 100 µg FP | 200 µg FP
Number analyzed (Participants) | 46 | 44 | 46 | 46 | 46
scores on a scale | 7.17 (2.912) | 5.54 (2.437) | 5.66 (2.280) | 5.29 (2.218) | 4.77 (2.433)
Statistical Analysis 1: Comparison: Placebo vs 25 µg FP; Test type: Superiority or Other; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-2.08 to -0.68], Standard Error of Mean 0.350 — Treatment difference (FP minus placebo) is presented as the difference in the adjusted means for treatment versus placebo
Statistical Analysis 2: Comparison: Placebo vs 50 µg FP; Test type: Superiority or Other; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-2.16 to -0.93], Standard Error of Mean 0.309 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs 100 µg FP; Test type: Superiority or Other; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-2.33 to -1.11], Standard Error of Mean 0.305 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs 200 µg FP; Test type: Superiority or Other; Mean Difference (Final Values) = -1.90, 95% CI 2-sided [-2.60 to -1.19], Standard Error of Mean 0.351 — Treatment difference is presented as the difference in the adjusted means for treatment versus placebo

2. Secondary Outcome: Weighted Mean Nasal Airflow at 2-5 Hours Post-dose (1-4 Hours Post-start of Challenge)
Description: Allergic rhinitis decreases the passage of air through the nose (nasal airflow) by increasing the nasal airway resistance. Rhinomanometry is used as an objective measurement of airway resistance. Nasal airflow was measured using active anterior rhinomanometry at pre-challenge, and then every 30 minutes from 0.5 to 4 hours post start of VCC. Weighted mean nasal airflow was calculated by dividing the value of the area under the response time curve between 1 and 4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each study period (Periods 1-4); up to Day 158
Population: All Subjects Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliters per second (mL/s)
Arm/Group | Placebo | 25 µg FP | 50 µg FP | 100 µg FP | 200 µg FP
Number analyzed (Participants) | 46 | 44 | 46 | 46 | 46
Milliliters per second (mL/s) | 335.20 (145.373) | 368.66 (144.230) | 375.94 (142.105) | 362.59 (142.216) | 411.65 (160.148)

3. Secondary Outcome: Weighted Mean Nasal Secretion at 2-5 Hours Post-dose (1-4 Hours Post-start of Challenge)
Description: Nasal secretion was measured by weighing tissues used by participants. Wet tissue weight assessments were made pre-challenge, and then every 30 minutes from 0.5 to 4 hours post start of challenge chamber throughout the study. Weighted mean nasal secretion was calculated by dividing the value of the area under the response time curve between 1 and 4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each study period (Periods 1-4); up to Day 158
Population: All Subjects Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: grams (g)
Arm/Group | Placebo | 25 µg FP | 50 µg FP | 100 µg FP | 200 µg FP
Number analyzed (Participants) | 46 | 44 | 46 | 46 | 46
grams (g) | 2.43 (2.203) | 1.63 (1.893) | 1.43 (1.458) | 1.26 (1.550) | 1.02 (1.271)

4. Secondary Outcome: Weighted Mean Eye Symptom Score at 2-5 Hours Post-dose (1-4 Hours Post-start of Challenge)
Description: The eye symptom score (total score of 0 [none] to 9 [severe]) was calculated as the sum of the symptom scores for watery eyes, itchy eyes, and red eyes, each of which was scored on a categorical scale from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), and was measured at pre-challenge, and then every 15 minutes from 0.25 to 4 hours post-start of challenge chamber. Weighted mean eye symptom score was calculated by dividing the value of the area under the response time curve between 1 and 4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each study period (Periods 1-4); up to Day 158
Population: All Subjects Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | 25 µg FP | 50 µg FP | 100 µg FP | 200 µg FP
Number analyzed (Participants) | 46 | 44 | 46 | 46 | 46
scores on a scale | 2.35 (2.240) | 1.52 (1.678) | 1.44 (1.711) | 1.93 (1.726) | 1.41 (1.491)

5. Secondary Outcome: Weighted Mean Global Symptom Score (GSS) at 5 Hours Post-dose (1-4 Hours Post-start of Challenge)
Description: GSS (total score=0-30) is calculated as the sum of sneeze, nasal itch, rhinorrhea, nasal obstruction, cough, itchy throat, itchy ears, watery eyes, itchy eyes, and red eyes SSs, each of which was scored on a categorical scale from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe), as was measured at pre-challenge, and then every 15 mins from 0.25 to 4 hours post-start of challenge chamber. Weighted mean global symptom score was evaluated by dividing the value of the area under the response time curve between 1 and 4 hours (calculated by trapezoidal rule) by the time interval of available data.
Time Frame: Day 8 of each study period (Periods 1-4); up to Day 158
Population: All Subjects Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | 25 µg FP | 50 µg FP | 100 µg FP | 200 µg FP
Number analyzed (Participants) | 46 | 44 | 46 | 46 | 46
scores on a scale | 11.14 (5.407) | 8.17 (4.302) | 8.24 (4.231) | 8.69 (4.346) | 7.13 (3.487)

6. Secondary Outcome: Glucocorticoid (GC) Receptor Biomarker Levels in Nasal Epithelial Scraping Samples: CCL2
Description: AROS Applied Biotechnology (AB) analyzed the nasal epithelial scrapings of participants and generated TaqMan (type of chemistry developed by AB to detect polymerase chain reaction [PCR] products) messenger ribonucleic acid (mRNA) biomarker expression data for CCL2, a steroid-responsive gene. Preliminary analysis of the mRNA abundance data was performed by Discovery Statistics. mRNA abundance data were normalized to the scores of GAPDH and 18S housekeeping genes. B-actin was not used. CCL2 data are presented by period to show the treatment-by-period interaction. ng, nanograms.
Time Frame: Day 1 (pre-dose) and Day 8 of each study period (Periods 1-4); up to Day 158
Population: All Subjects Population. The data presented for each period are an average of the data collected on Day 1 and Day 8 of each period. Only those participants contributing data at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Copies of RNA detected per 50ng of total
Arm/Group | Placebo | 25 µg FP | 50 µg FP | 100 µg FP | 200 µg FP
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Copies of RNA detected per 50ng of total
  Period 1, n=12, 12, 12, 11, 11 | 12396.08096 [5928.406 to 25919.75529] | 1377.248941 [678.7116 to 2794.728503] | 1231.251053 [605.7205 to 2502.769902] | 3340.460181 [1599.611 to 6975.866146] | 3377.403394 [1625.327 to 7018.188693]
  Period 2, n=11, 11, 11, 12, 11 | 4206.320679 [1991.881 to 8882.624596] | 2192.232108 [1015.906 to 4730.634081] | 1765.627412 [849.2589 to 3670.781431] | 2342.488506 [1127.738 to 4865.715164] | 2821.11204 [1355.137 to 5872.967075]
  Period 3, n=11, 11, 11, 12, 12 | 4135.167835 [1987.132 to 8605.171059] | 3612.444351 [1730.839 to 7539.553498] | 2184.76185 [1051.383 to 4539.910315] | 1229.316666 [609.3241 to 2480.157112] | 2505.03196 [1234.885 to 5081.594294]
  Period 4, n=12, 11, 11, 11, 12 | 10111.38124 [5019.348 to 20369.18487] | 3523.276415 [1674.529 to 7413.114228] | 2615.352938 [1249.52 to 5474.157686] | 1917.918706 [889.5355 to 4135.205377] | 1071.598621 [515.8547 to 2226.060108]

7. Secondary Outcome: Glucocorticoid (GC) Receptor Biomarker Levels in Nasal Epithelial Scraping Samples: 18S, B-actin, DUSP_1_T1, FKBP5, GAPDH, GILZ, PLAU, PTGS2, and RGS2
Description: AROS Applied Biotechnology (AB) analyzed the nasal epithelial scrapings of participants and generated TaqMan (type of chemistry developed by AB to detect polymerase chain reaction [PCR] products) messenger ribonucleic acid (mRNA) biomarker expression data for 7 steroid-responsive genes (DUSP_1_TI, FKBP5, GILZ, PLAU, CCL2, PTGS2, and RGS2) and 3 housekeeping reference genes (GAPDH, 18S, and b-actin). Preliminary analysis of the mRNA abundance data was performed by Discovery Statistics. mRNA abundance data were normalized to the scores of GAPDH and 18S housekeeping genes. B-actin was not used.
Time Frame: Day 1 (pre-dose) and Day 8 of each study period (Periods 1-4); up to Day 158
Population: All Subjects Population. The data presented are an average of the data collected on Day 1 and Day 8 of each treatment period. Only those participants contributing data at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: RNA copies detected per 50 ng total RNA
Arm/Group | Placebo | 25 µg FP | 50 µg FP | 100 µg FP | 200 µg FP
Number analyzed (Participants) | 46 | 45 | 45 | 46 | 46
RNA copies detected per 50 ng total RNA
  18S | 6439292568 [5953473924 to 6964755253] | 6109603485 [5653823536 to 6602125890] | 5822423622 [5388052053 to 6291813164] | 6218835383 [5759650434 to 6714628599] | 6222906532 [5758553637 to 6724703483]
  B-actin | 1978137.142 [1761487.822 to 2221432.646] | 1481307.983 [1316851.063 to 1666303.352] | 1629006.342 [1448708.283 to 1831743.28] | 1630387.679 [1451329.134 to 1831537.671] | 1543748.32 [1374839.809 to 1733408.402]
  DUSP_1_T1 | 107004.8077 [87973.18828 to 130153.6195] | 104633.517 [85852.10596 to 127523.6379] | 107031.4158 [88881.02888 to 128888.2916] | 118158.2593 [97226.90284 to 143595.7933] | 113323.9632 [91653.05005 to 140118.8573]
  FKBP5 | 28739.3975 [24256.97193 to 34050.12675] | 155791.0745 [131185.2632 to 185012.0837] | 174963.5715 [147311.3952 to 207806.4043] | 177935.1307 [150181.7514 to 210817.2961] | 151362.3934 [127521.6515 to 179660.2684]
  GAPDH | 5776051.293 [5326118.123 to 6263993.356] | 6143058.472 [5659602.91 to 6667811.859] | 6451580.253 [5943884.286 to 7002640.993] | 6008446.351 [5540570.46 to 6515832.227] | 5972472.493 [5507396.953 to 6476821.624]
  GILZ | 13601.9459 [11833.92763 to 15634.1105] | 26629.75763 [23090.34785 to 30711.70672] | 29304.22353 [25490.27435 to 33688.8299] | 28832.53255 [25122.37093 to 33090.62412] | 27304.24721 [23763.4653 to 31372.60943]
  PLAU | 26364.53138 [22020.16973 to 31565.99261] | 18550.2079 [15417.62826 to 22319.27033] | 18810.56868 [15681.73421 to 22563.67116] | 20918.214 [17454.94721 to 25068.63365] | 21692.66346 [18117.03777 to 25973.98394]
  PTGS2 | 42479.35246 [34135.93482 to 52862.04685] | 31120.01509 [24904.20116 to 38887.22762] | 35049.7556 [28101.49486 to 43716.01489] | 38443.85612 [30827.02769 to 47942.67187] | 33657.71928 [27031.4341 to 41908.32284]
  RGS2 | 55084.11432 [45323.01163 to 66947.44108] | 45255.7763 [37098.26279 to 55207.04028] | 54186.44212 [44490.27052 to 65995.78907] | 50507.30739 [41546.43595 to 61400.88895] | 50373.91657 [41440.13318 to 61233.67074]

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were collected in the 46 participants who received placebo and FP 25, 50, and 100 µg treatments, and in the 47 participants who received FP 200 µg.
Arm/Group | Placebo | 25 µg FP | 50 µg FP | 100 µg FP | 200 µg FP
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/46 | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 4/46 | 6/46 | 3/46 | 2/46 | 1/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=46) | 25 µg FP (N=46) | 50 µg FP (N=46) | 100 µg FP (N=46) | 200 µg FP (N=47)
Nasopharygitis (Infections and infestations) | 1 | 2 | 0 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.